CLINICAL TRIAL: NCT04144582
Title: Multiple-center, Single-arm, Phase II Study on Sintilimab Combined With Docetaxel in Non-driver Gene Mutation Advanced NSCLC Patients Who Had Failed With Double Platinum-based Chemotherapy
Brief Title: Sintilimab Combined With Docetaxel for Standard Chemotherapy Failure Non-driver Gene Mutation Metastatic Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yongchang Zhang (Other)
Responsible Party: Sponsor-Investigator, Yongchang Zhang, Professor, Hunan Province Tumor Hospital
Organization: Hunan Province Tumor Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STORM
Record Dates: First submitted 2019-10-28; First posted 2019-10-30 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-03

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sintilimab Combined With Docetaxel (Experimental): Sintilimab Combined With Docetaxel for Metastatic or Non-driver Gene Mutation Non-small Cell Lung Cancer
  Interventions: Drug: Sintilimab Combined With Docetaxel Monotherapy

INTERVENTIONS:
Drug: Sintilimab Combined With Docetaxel Monotherapy — Sintilimab 200mg i.v q3w , Docetaxel 75mg/m2 i.v q3w

SUMMARY:
The purpose of this study is to assess the safety and effectiveness of Sintilimab Combined With Docetaxel in Non-driver Gene Mutation NSCLC patients who failed with double platinum-based chemotherapy

ELIGIBILITY:
Inclusion Criteria:

* Life expectancy exceeds 3 months
* The investigator confirmed at least one measurable lesion according to the RECIST 1.1 standard.

Exclusion Criteria:

* small cell lung cancer or small cell lung cancer
* Currently involved in interventional clinical research or treatment, or have received other research drugs or used research equipment within 4 weeks prior to the first dose;
* Previously received the following treatments: anti-PD-1, anti-PD-L1 or anti-PD-L2 drugs or drugs that stimulate or synergistically inhibit T cell receptors (eg, CTLA-4, OX-40, CD137);

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
ORR | Approximately 1 years
  To measure the patients's overall response rate

SECONDARY OUTCOMES:
PFS | Approximately 1 years
  Progression free survival
OS | Approximately 1 years
  Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Yongchang Z MD, MD, Principal Investigator — Hunan Province Tumor Hospital
Locations (2):
- China (2):
  - Hunan Provincal Tumor Hospital, Changsha, Hunan
  - Yongchang Z MD, Changsha, Hunan